CLINICAL TRIAL: NCT03304561
Title: Contralateral Strength Training Effects on Functional Outcomes in Patients Who Had Undergone ACL Reconstruction: Randomized Controlled Trial
Brief Title: The Effect of Contralateral Limb Training on Functional Outcomes in Patients With ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, GULCAN HARPUT, Phd, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: knee; rehabilitation; ACL; Contralateral training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional rehabilitation (Experimental): patients in this groups is going to recieve traditional rehabilitation programme for 3 months after ACL recontsruction
  Interventions: Other: Traditional rehabilitation
- Cross-over training (Experimental): patients in this programme is going to recieve isokinetic exercise programme targeting unilvolved limb during rehabilitation. for the first 4 weeks after ACL reconstruction traditional rehabiitation programme is going to applied to the subjects. after 4 weeks, isokinetic strenghtening programme at 60˚/second angular velocity, between 0-90 degree knee flexion until 3 months after ACL reconstructon
  Interventions: Other: Cross-over training

INTERVENTIONS:
Other: Traditional rehabilitation — traditional ACL rehabilitation program
  Other Names: Standard post-operative ACL rehabilidation program
  Arms: traditional rehabilitation
Other: Cross-over training — Cross-over training addition to the traditional rehabilidation
  Arms: Cross-over training

SUMMARY:
Quadriceps and hamstring muscle strenghts have important role in returning to sport after ACL reconstruction and one of the main focus of rehabilitation is to improve strenght of these muscles. With the strenghtening of the contralateral limb (cross-over training) we aimed to improve the strenght of the quadriceps

DETAILED DESCRIPTION:
Returning to sport after ACL reconstruction is not at desired level among athletes. Quadriceps and hamstring muscle strenghts have important role in returning to sport after ACL reconstruction. Cross-over training is recomended during rehabilitation after ACL reconstrucion. Yet duration of the training, frequancy and type of exercise interention are not clear for the cross-over training. Ain of the study is to investigate the effects of cross-over training on muscle strenght

ELIGIBILITY:
Inclusion Criteria:

* having surgery of ACL reconstruction on one side
* having no problem at least six month on the nonsrgical side
* recieving the rehabilitation programme at hacettepe university, physiotherapy department

Exclusion Criteria:

* refusing to include to the study
* having revision ACL surgery
* addition of PCL or cartilage surgery addition to the ACL surgery
* not participating to the rehabilidation program regularly over 3 month after sugery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
quadriceps and hamstring muscle strenght | 6 month
  quadriceps strength change during the first, second and sixth months of the rehabilitation proccess after ACL reconstruction surgery. the strength measurements will conducted on isokinetic dynamometer (isomed 2000)

SECONDARY OUTCOMES:
functional outcomes | 6 month
  one leg hop test, vertical jump test on the sixth month after surgery. the functional outcomes will be measured only at the sixth month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: volga tunay, PhD, Study Director — volgamel@yahoo.com
Locations (1):
- Sports Physiotherapy Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No